CLINICAL TRIAL: NCT04909008
Title: Exercise Training to Improve Pulmonary Haemodynamic and Right Ventricular Function in Heart Failure Patients With Pulmonary Hypertension
Brief Title: Exercise Training to Improve Cardiopulmonary Hemodynamics in Heart Failure Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Mayo Clinic (Other)
Collaborators: Florida Heart Research Institute (Other)
Responsible Party: Principal Investigator, Bryan Taylor, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-011347
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2025-04-21 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Pulmonary Hypertension
Keywords: Exercise training; Right ventricle; Exercise capacity; Quality of life
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training (Experimental): Two sets of exercise testing (before and after) 10 weeks of supervised exercise training (3 sessions per week) at Mayo Clinic Florida.
  Interventions: Other: Exercise Training
- Control Groups (No Intervention): Two sets of exercise testing while continuing with standard medical care in between.

INTERVENTIONS:
Other: Exercise Training — 10 weeks of supervised exercise training, 3 sessions per week at the cardiac rehab clinic at Mayo Clinic Florida.
  Other Names: Cardiac Rehab
  Arms: Exercise Training

SUMMARY:
This research study is being done to find out if exercise therapy can help improve the heart function, overall health, and quality of life of patients with pulmonary hypertension caused by heart failure.

DETAILED DESCRIPTION:
The purpose of this research is to see if taking part in structured exercise training will improve the ability to exercise, the function of the heart, and the function of the blood vessels that supply the lungs in patients with heart failure and pulmonary hypertension. After enrollment all patients will complete exercise testing. Patients will be randomized to either 10 weeks of exercise training (3 times per week) or will continue standard medical care. All patients will undergo detailed exercise testing before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* NYHA functional class I-IIIb.
* LVEF < 40%.
* Clinically-stable for > 3 months [no change in disease status or medication].
* Willing and able to provide written informed consent and perform cycle-ergometer or treadmill based exercise.

Exclusion Criteria:

* NYHA class IV HF.
* Diagnosis of diastolic HF.
* Comorbidities such as obesity (BMI >36), uncontrolled systemic hypertension, type 2 diabetes, and COPD (FEV1 <50%).
* Musculoskeletal or other conditions that would limit exercise participation.
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2max) measured in mL/kg/min | 10 weeks
  VO2max is the maximal measured oxygen uptake during a symptom limited exercise test.

SECONDARY OUTCOMES:
Mean pulmonary arterial pressure (mPAP) measured in mmHg | 10 weeks
  mPAP will be measured at rest and during exercise and is a measure of pulmonary vascular pressure.
Pulmonary vascular resistance (PVR) measured in dynes | 10 weeks
  PVR will be measured at rest and during exercise and is a measure of pulmonary hemodynamic function.
Right ventricular contractile function measured as % fractional area change (RV FAC). | 10 weeks
  RV FAC is a measure of overall contractile function of the right ventricle.
Left ventricular contractile function measured as % fractional area change (LV FAC). | 10 weeks
  LV FAC is a measure of overall contractile function of the left ventricle.
Slope of the relationship between mean pulmonary arterial pressure and cardiac output (mPAP-Q slope) measured in mmHg/L/min. | 10 weeks
  The mPAP-Q slope during exercise is a measure of the pulmonary hemodynamic response to exercise. A slope >3 is 'abnormal', and a steeper slope is related to poorer pulmonary hemodynamic function.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan J Taylor, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials